## **Addressing Obesity in Early Care and Education Settings**

NCT04140032

December 17, 2024



Addressing Childhood Obesity in Early Care and Education Settings UCLA Center for Cancer Prevention and Control Research and Child Care Resource Center

## **Table of Contents**

| Abbreviations | 4 |
|---|---|
| Project Personnel | 4 |
| Proposed Project Timeline | 5 |
| Proposed Data Collection Timeline | 5 |
| Data Collection Timeline Modifications from Cohort 1 | 5 |
| Data Collection Timeline Modifications due to COVID-19 | 6 |
| Project Phases | 6 |
| Phase I: Recruitment | 7 |
| Recruitment Flow Sheet | 7 |
| Recruitment of Sites Cohort 1 | 7 |
| Recruitment of Sites Modifications from Cohort 1 | 8 |
| Recruitment of Sites Modifications due to COVID-19 | 8 |
| Recruitment of Sites Cohort 3 | 8 |
| Initial Recruitment Call | 8 |
| Initial Recruitment Call Modifications from Cohort 1: | 8 |
| In-Person Meeting 1 | 9 |
| In-Person Meeting 1 Planned Modifications from Cohort 1 | 9 |
| In-Person Meeting 1 Modifications due to COVID-19 | 9 |
| Site Demographics Data Collection Meeting | 9 |
| Site Demographics Collection Meeting Modifications due to COVID-19 | 9 |
| Phase II: Baseline Data Collection | 10 |
| Site Director Survey Distribution and Collection | 10 |
| Site Director Survey Distribution and Collection Modifications due to COVID-19 | 10 |
| Teacher Survey Distribution and Collection | 10 |
| Teacher Survey Distribution and Collection Modifications due to COVID-19 | 10 |
| Teacher Survey Distribution and Collection Modifications due to COVID-19 | 11 |
| Parent Survey Distribution and Collection | 11 |
| Parent Survey Distribution and Collection Modifications due to COVID-19 | 11 |
| Survey Reminder Emails | 12 |
| Parent On-site Recruitment/ Tabling Events Cohort 1 Data Collection: | 13 |
| Pilot Testing Parent Survey Procedure | 13 |
| Survey Entry | 13 |

| Unique IDs | 13 |
|------------------------------------------------------------------|----|
| Unique ID Modifications due to COVID-19 | 14 |
| Site Director Survey Entry | 14 |
| Teacher Survey Entry | 14 |
| Parent Survey Entry | 14 |
| EPAO | 15 |
| EPAO Modifications due to COVID-19 | 15 |
| Height and Weight Measurements | 15 |
| Height and Weight Modifications due to COVID-19 | 16 |
| Gift Cards | 16 |
| Gift Card Amounts | 17 |
| Phase III: Randomization and Implementation | 17 |
| Randomization of Sites | 17 |
| Implementation | 18 |
| Implementation Tracking | 18 |
| Coaching | 19 |
| Coaching Modifications due to COVID-19 | 19 |
| Family Child Care (FCC) Coaching – Cohort 2 | 20 |
| Coaching Data Entry | 20 |
| Parent Engagement | 20 |
| Parent Engagement Modifications due to COVID-19 | 20 |
| Parent Website | 20 |
| Phase IV: Follow-up Data Collection | 21 |
| Follow-Up Data Collection | 21 |
| Cohort 1 Follow-up Data Collection Modifications due to COVID-19 | 21 |
| Cohort 2 Data Collection Modifications due to COVID-19 | 21 |
| Follow-up Surveys | 21 |
| Paper Follow-up Surveys | 21 |
| Electronic Follow-Up Surveys- Cohort 1 Follow-up | 22 |
| Follow-up EPAO | 22 |
| Follow-up Height and Weight | 22 |
| Phase V: Evaluation | 23 |
| Program Evaluation | 23 |
| Process Evaluation | 23 |
| Outcome Evaluation | 23 |
| APPENDIX I: Initial Director Call Talking Points | 24 |

| APPENDIX II: Initial Call | 25 |
|-------------------------------------------------|----|
| APPENDIX III: In-Person Meeting 1 | 26 |
| APPENDIX IV: Participant Survey Packets | 27 |
| APPENDIX V: How to Enter Preschool Project Data | 28 |
| APPENDIX VI: How to Generate a Unique ID | 30 |
| APPENDIX VII: EPAO | 32 |
| APPENDIX VIII: Height and Weight Materials | 33 |
| APPENDIX IX: Scale Calibration Summary | 34 |

#### BOX SEARCH TERMS ARE BOLD, UNDERLINED, AND ITALICIZED THROUGHOUT DOCUMENT

## **Abbreviations**

CACFP – Child and Adult Care Food Program (a.k.a. the food program)

CCRC – Child Care Resource Center

CPCR – Cancer Prevention and Control Research Center (at UCLA)

EPAO – Environment and Policy Assessment and Observation (observation tool)

FCC – Family Child Care home/provider

H&W – Height and Weight

NAPSACC – Nutrition and Physical Activity Self-Assessment for Child Care (Site Director survey)

## Project Personnel

| UCLA:CCRC:Roshan Bastani - Primary Investigator (PI)Ana (Lily) Duarte - Supervisor, Coaching, Resource and ReferralCindy Chang - Senior StatisticianBrianna Briones - Senior Research Analyst, Research andPaul Chung - PIEvaluationJennie Coleman - Project CoordinatorAdriana Garcia - Coach, Resource and Referral |
|---|
| Cindy Chang – Senior Statistician Brianna Briones – Senior Research Analyst, Research and Evaluation |
| Paul Chung – PI Evaluation |
| č |
| Jennie Coleman - Project Coordinator Adriana Garcia – Coach, Resource and Referral |
| Burt Cowgill - Co-Investigator Elizabeth (Liz) Melendrez - Manager, Resource and Referral |
| Kate Crespi – Statistician Jared Nineberg – Senior GIS Analyst, Research and Evaluation |
| Mayte Cruz - Project Staff (2019- Aug 2020) Olivia Pillado - Manager, Research and Evaluation |
| Beth Glenn - Co-Investigator Cynthia Renteria - Assistant Director, Resource and Referral |
| Michelle Guerra – Field Staff (2019- Aug 2020) Susan Savage - Director, Research and Evaluation |
| Alison Herrmann - Co-Investigator Cyndi Trujillo –Manager, Resource and Referral |
| Lindsay du Plessis – Research Scientist |
| Chris Johansen - Post-Doc Fellow <u>UCLA Interns</u> : |
| Varduhi Niksalyan – Project Staff (2020 – Aug 2021) Roline Dahl – undergraduate intern (2019-2020) |
| Alexandra Nordyke – Project Assistant (Aug 2020- Celeste Martinez – undergraduate intern (2019-2020) |
| present) |
| Bernadett Leggis – Field Staff Mominah Subhan – undergraduate intern (2019-2020) |
| Vincent Liu – Project Assistant (2019-Aug 2020) Ayushi Bommireddipalli – undergraduate intern (2021 - present) |
| Jessica Richardson – Field Staff (2019-2020) |
| Maria Santos – Project Staff (Sept 2020 – July 2021) |
| Djosy Charles – Project Staff (Feb 2021 – Oct 2021) |
| Diana Trujillo – Project Staff (Aug 2021 – present) |

## Protocol

NIH R01 Clinical Trial R01HD091136.

UCLA IRB approval number: 19-000570-CR-00002.

The purpose of this protocol is to guide the recruitment of sites/participants and implementation of program activities for University of California-Los Angeles (UCLA) and Child Care Resource Center (CCRC)'s A-B-C Healthy Me/Soy Saludable Project to Address[ing] Obesity in Early Care and Education Settings.

This project will recruit preschools from LA County's San Fernando Valley, Santa Clarita Valley, and Antelope Valley, specifically targeting preschools in low to medium-income zip codes. Three cohorts of 20 schools (n=60) over three instructional years (~Sept 1 – June 30) will be recruited and randomized (10 intervention; 10 control/delayed intervention per year).

Program activities were designed in line with the Healthy-by-Default framework and include the following:

- Integration of Sesame Street Healthy Habits for Life curriculum
- Teacher and site director coaching
- Nutrition and physical activity policy support including family-style meals and healthy celebrations
- Parent engagement sessions
- Implementation Activity Table (word doc):Box Project misc.-->Research Plan Component Table\_Preschool Policy, Teacher, Parent Activities

## **Proposed Project Timeline**

Cohort 1: September 2019-June 2020

Cohort 2: May 2020-June 2021 Cohort 3: May 2021-June 2022

Follow-up (post) surveys will occur immediately after intervention completion each year.

## Proposed Data Collection Timeline

| Week 1 | Week 2 | Week 3 | Week 4 | Week 5 | Week 6 | Week 7 |
|---|---|---|---|---|---|---|
| Initial Recruitm | ent Call/Email fro | m CCRC | | | | |
| In-person Meeting with Site, CCRC, and UCLA | | | | | | |
| Site director and teacher surveys | | | | | | |
| | | EPAO Observations | | | | |
| | | Parent Recruitment | | | | |
| | | Height and Weight Measurements | | | nts | |

#### Data Collection Timeline Modifications from Cohort 1

The proposed data collection timeline has been updated from cohort 1. The cohort 1 data collection strategy was staggered by participant pool; the site director survey was delivered and collected a week later. At collection, the teacher surveys were delivered and collected a week later or at EPAO. At teacher survey collection, parent surveys were delivered and left with site staff to distribute. We originally structured recruitment this way as to not overwhelm the site and to give the director time to digest the program and complete site level data before engaging teachers. However, after meeting with site directors in cohort 1, we realized that this staggering pushed recruitment back by at least 3 weeks. By combining the site director and teacher survey distribution in cohort 2, we will be able to more efficiently collect site director and teacher data thus allowing more time for the intervention.

## Data Collection Timeline Modifications due to COVID-19 Data Collection Timeline Modifications due to COVID-19—Cohort 1 Follow-up and Cohort 2 baseline

Due to COVID-19, all participant surveys for cohort 1 follow-up and cohort 2 baseline will be available online via Qualtrics; paper surveys will be available to those sites that do not communicate with parents via email. All participants will need to provide an email for us to provide them directly with the survey link and their unique password. In order to protect the privacy of each survey, UCLA will have to pre-assign an ID and password to each participant. The link and unique password will then be emailed to each participant at the email provided by the site.

Email addresses were collected from the site. An opt-out model was used to notify site participants of the program and that their email will be shared with UCLA for more information on participation. A flyer with this information was given to the site director to distribute to parents. After a week to review/notify with parents, UCLA would ask the site director to provide parent and teacher emails that the site has on file. If a parent or teacher verbally opted out, their email will not be shared.

Paper surveys were also delivered to all sites. Some sites only returned paper surveys and 2 sites did not collect parent emails but went straight to paper.

Additionally, the EPAO will not be conducted as long as social distancing orders are in effect.

#### Data Collection Timeline Modifications— Cohort 2 Follow-up and Cohort 3 baseline

Majority of Cohort 2 sites preferred paper and the paper response rate was better for all sites, starting 5/25/21(cohort 2 follow-up) all data collection will be conducted via paper only.

## **Project Phases**

Phase I: Recruitment

Phase II: Baseline Data Collection

Phase III: Randomization and Implementation

Phase IV: Follow-up Data Collection

Phase V: Evaluation

## Phase I: Recruitment

## Recruitment Flow Sheet



#### Recruitment of Sites Cohort 1

CCRC provided UCLA with a list of center-based preschools in their network, which are in low to middle-income zip codes in the San Fernando Valley. Additional information included: location, size (i.e., capacity) and CACFP participation.

UCLA then randomized the list for CCRC to contact.

Centers must have more than 20 preschool aged children (2-5 years old) enrolled. The schools that participated in the formative data collection were contacted first. If a school was unable or unwilling to participate, that it is noted, and another site is contacted for recruitment.

For sites that decline initial participation, we will determine if they would be interested in participating in future years. A deferred list of sites will be maintained for contact in the next program year.

For cohort 1, recruitment began September 9, 2019. For cohort 2, recruitment began May 20, 2020. For cohort 3, recruitment began April 19, 2021.

#### Recruitment of Sites Modifications from Cohort 1

Since CCRC provided UCLA with a provider list during cohort 1, all centers not contacted during cohort 1 were added to the cohort 2 contact list. Additionally, Centers in the Santa Clarita and Antelope Valleys were included. Age range was expanded to include 2-6 years old since siblings may be in the same classroom due to COVID-19. Zip code income was dropped as a stratifying variable.

The cohort 2 contact list was broken down into three recruitment rounds: 1) centers that 'deferred year 1' and 'CACFP participants', 2) centers that receive CCRC subsidy but non-CACFP'; and 3) 'unsubsidized, non-CACFP'. CCRC contacted schools from this list.

Family Child Care (FCC) providers were included in cohort 2 as a pilot for this population. FCCs should have a minimum of 6 eligible participants. 4 FCCs were recruited in cohort 2.

See APPENDIX I: Initial Director Call Talking Points for more information on what to bring to the initial call and talking points.

#### Recruitment of Sites Modifications due to COVID-19

Additionally, with widespread preschool closures due to COVID-19, we decided to offer our control sites from cohort 1 the opportunity to convert into intervention sites for cohort 2. This offer was extended to the cohort 2 control sites as well. Control sites were added back into the recruitment pool to confirm interest in another year of participation. Due to low participation during follow-up data collection (August 2021) at the cohort 2 control sites, these sites did not convert to cohort 3 intervention sites, but instead received coaching every other month.

#### Recruitment of Sites Cohort 3

Deferred cohort 2 sites were contacted first for cohort 3 (~n=54). Once CCRC contacted all schools on the deferred list, CCRC pulled from the original list for additional centers not yet contacted.

#### Initial Recruitment Call

CCRC contacted the identified schools via phone to recruit and answer questions. CCRC initially sent an interest email to the site directors explaining the study, its components, and the expectations of each site. Within the next few days, CCRC followed up the email with a phone call to discuss the program. Interested sites then scheduled an in-person meeting.

#### See APPENDIX II: Initial Recruitment Call for what to bring for Initial Recruitment Call

#### Initial Recruitment Call Modifications from Cohort 1:

For cohort 2, we began with an initial call rather than an email since it took multiple attempts to connect with site directors, as many site directors reported not getting the email or asked it to be re-sent after the initial call. In cohort 1, many sites agreed to the in-person meeting after the initial call. However, we understand that some sites will require follow-up calls to confirm interest since they often take this information back to their owners/ teachers. Follow-up calls are scheduled during the initial call to ensure the site director's availability. We believe condensing this recruitment step will allow us to enroll sites more efficiently.

## After Site Agrees to Participate

## In-Person Meeting 1

The purpose of an in-person meeting 1 is to meet with the site to review the project, address any site questions or concerns, and enroll interested sites in participation. The in-person meeting 1 is scheduled during the initial call, and communication is documented in the initial call log. We encourage site directors to review all materials with teachers to ensure teacher buy-in.

Program activities and logistics are discussed at the in-person meeting 1. If a site is interested, a second data meeting is scheduled a week later with UCLA staff to collect site demographics and the site director survey is given to site director. A week later, the director survey is collected, and the teacher surveys are delivered.

#### See APPENDIX III: In-Person Meeting 1 for what to bring for In-person Meeting 1

#### In-Person Meeting 1 Planned Modifications from Cohort 1

For cohort 2, we plan to deliver the site director and teacher surveys at the first in-person meeting. At this time, we will also schedule the EPAO for 1-2 weeks from the in-person meeting. By scheduling the EPAO at the first in-person meeting, we are setting a stricter timeline for data collection, since the EPAO is to be done within 2 weeks of enrollment. During the in-person meeting, we will also discuss each data collection activity and outline site specific plans for how to deliver each survey efficiently to their participation pool. At the EPAO, we will collect the site director and teacher surveys as well as deliver the parent surveys. At some sites, we may be able to collect teacher and site director surveys and deliver parent surveys in between the first in-person meeting and the EPAO; if we are able to do so, this will allow for more time to recruit parents. Condensing the survey delivery into one visit will allow us to collect data more efficiently as well as limit interference with site activities.

### In-Person Meeting 1 Modifications due to COVID-19 Cohorts 2 and 3

Due to COVID-19, the first in-person meetings for Cohorts 2 and 3 are held via Zoom. UCLA and CCRC will meet with the site director to review the <u>RECRUITMENT POWERPOINT</u> and answer any questions. If the site director would like to enroll, UCLA will then schedule a data collection meeting within the next week to collect site demographics.

Follow-up in-person meeting 1 with an email to the site director containing: 1) Calendar invite for site demographics data collection meeting, 2) Director and teacher participation letters, 3) Participation agreement, and 4) List of policy documents to submit.

## Site Demographics Data Collection Meeting

After a site agrees to participate, a follow-up meeting to collect basic site demographics and finalize the data collection plan with UCLA is scheduled. The purpose of this meeting is for UCLA to collect baseline demographic information about the site (i.e. Enrollment numbers, food patterns, CACFP/menu guidelines, etc....) and discuss how best to collect data from the site. Data is logged in the Site Demographics excel sheet on Box.

Site Demographics Collection Meeting Modifications due to COVID-19
Site Demographics Collection Meeting Modifications - Cohorts 2 and 3

Due to COVID-19, data collection meetings for cohorts 2 and 3 were conducted via Zoom instead of in-person. UCLA staff uses the *ABC HEALTH ME INTRODUCTION DATA POWERPOINT* to help guide the meeting.

## Phase II: Baseline Data Collection

## 1) Survey Collection

Cohort 1 Baseline survey collection began 9/18/21 (conducted via paper)

Cohort 1 Follow-up survey collection began 7/8/20:

Data collection for Cohort 1 Follow-up sites was conducted electronically. Two Cohort 1 Control sites converted to Cohort 2 intervention sites. These 2 "converted" sites requested data collection to be conducted via paper.

Cohort 2 Baseline survey collection began 9/15/2020

Data collection for Cohort 2 baseline survey was conducted via paper and electronically (protocols below). Cohort 2 sites could request data collection to be conducted via paper in addition to electronically.

Cohort 2 Follow-up survey collection began 5/25/2021 (conducted via paper)

Cohort 3 Baseline survey collection began 9/29/2021 (conducted via paper)

### Site Director Survey Distribution and Collection

Director surveys is an abridged version of NAPSACC (gonapsacc.com). The site director should receive a paper survey at the first in-person meeting and should return the survey to UCLA at the next site visit.

#### See APPENDIX IV: Participant Survey Packets

Site Director Survey Distribution and Collection Modifications due to COVID-19 Cohort 1 Follow-up and Cohort 2 Baseline Data collection:

Due to COVID-19, in-person data collection paused, leaving surveys to be distributed electronically. After the first in-person meeting, UCLA will email the site director with the survey link and unique password. All **SURVEY LINKS** are on Box.

Paper versions were delivered to site directors who preferred paper or did not complete online.

Site Director Survey Distribution and Collection Modifications – Cohort 2 Follow-up and Cohort 3 Baseline

Since majority of site directors preferred paper, paper will be the primary survey collection mode moving forward. For cohort 2 follow-up and cohort 3, data collection will be conducted via paper only.

## Teacher Survey Distribution and Collection

Teacher materials should be delivered at the same time as or when picking up the site director survey. The site director will act as the primary conduit for teacher communication. Teachers will submit completed surveys in a sealed envelope to the site director for UCLA collection. The site director will keep the sealed surveys in a locked cabinet until UCLA staff picks them up.

#### **See APPENDIX IV: Participant Survey Packets**

Teacher Survey Distribution and Collection Modifications due to COVID-19 Cohort 1 Follow-up and Cohort 2 Baseline

Due to COVID-19, in-person data collection paused, leaving surveys to be distributed electronically. All <u>SURVEY</u> <u>LINKS</u> are on Box. In order to protect the privacy of each electronic survey, UCLA staff will have to pre-assign an ID and password to each participant. The link and unique password will then be emailed to each participant. Paper surveys can be provided to sites that prefer.

Teacher emails must be collected from the site in order to provide teachers with a survey link and unique password. A <u>TEACHER EMAIL COLLECTION FLYER</u> sheet will be emailed to the site director to provide to the teachers. The flyer provides information about the program and explains the opt-out model of email collection. If a teacher does not want to participate, they are told to let their director know. After a week, UCLA will reach out to collect teacher emails from the director.

Once teacher emails have been collected, UCLA will send each teacher the <u>TEACHER BASELINE SURVEY LINK</u>

AND PASSWORD EMAIL explaining the program as well as providing the survey link and password.

Since the online priority was parent enrollment, teacher emails were collected after parent emails. Some sites chose to do paper surveys with their teachers.

Depending on the response rate, UCLA paper surveys may be delivered to sites in order to increase participation. During Cohort 2 baseline data collection, most teachers preferred paper surveys. Beginning 10/19/20, paper surveys were the primary survey collection method.

## Teacher Survey Distribution and Collection Modifications due to COVID-19 Cohort 2 Follow-up and Cohort 3

During Cohort 2 baseline data collection, most teachers preferred paper surveys. Cohort 2 follow-up and cohort 3 data collection will be conducted via paper only.

## Parent Survey Distribution and Collection

Parent surveys and consent forms are delivered in envelopes to the site and distributed by teachers in their classrooms. Some sites elect to have the director hand out the surveys to parents directly. Parent materials are provided to teachers during EPAO to hand out to their parents. UCLA staff should discuss the distribution process with teachers and/or the site director before leaving the surveys (e.g. Put parent surveys in cubbies during naptime or slip envelopes with child's name into sign out log.) Additional surveys can be delivered if the site needs more copies. The <u>PARENT</u> <u>NOTIFICATION FLYER</u> is available for sites who would like to let parents know to keep an eye out for what's to come.

Teachers turn in all submitted parent envelopes to the site director to keep in a locked cabinet until pick-up by UCLA staff. Materials are *collected weekly*. UCLA staff delivers gift cards within 48 hours if not on the same day. Due to shipping delays, gift cards are scheduled for delivery within 48 hours of UCLA project staff receiving gift cards.

#### See APPENDIX IV: Participant Survey Packets

## Parent Survey Distribution and Collection Modifications due to COVID-19 Cohort 1 Follow-up and Cohort 2 Baseline

Due to COVID-19, in-person data collection has been paused for Cohort 1 Follow-up and Cohort 2 Baseline, leaving surveys to be distributed electronically. All <u>SURVEY LINKS</u> are on Box. In order to protect the privacy of each electronic survey, UCLA staff will have to pre-assign an ID and password to each participant. The link and unique password will then be emailed to each participant. Paper surveys were delivered to sites that do not communicate via email with parents or do not believe their parents will participate electronically.

Parent emails must be collected from the site in order to provide parents with the survey link and unique password. A <u>PARENT EMAIL COLLECTION FLYER</u> and <u>PARENT EMAIL COLLECTION TEMPLATE</u> will be emailed to the site director to email to their parents. The flyer provides information about the program and explains the opt-out model of email collection. If a parent does not want to participate, they are told to let their site director know. After a week, UCLA staff will reach out to collect parent emails from the site director.

Once parent emails have been collected, UCLA staff will send each parent the <u>PARENT BASELINE SURVEY LINK</u>
<u>AND PASSWORD</u> email explaining the program and providing the survey link and password. Email addresses and unique survey information will be extracted from our Unique ID tacking data and compiled using a Python code. Emails will be

sent to participating parents via the webhost MailChimp. The email will contain a link to the survey as well as a required password to enter the survey. The link and password will be assigned to their unique ID.

In the event of two emails provided for one child, we will send the first email to the mother. If we cannot discern which email belongs to the child's mother, we will send the emails to the first email address listed alphabetically. If we have trouble contacting a family with two emails, we may send follow-up emails to the second provided address.

In the event of one parent having two or more children participating in the study, we will use a different email template and provide the passwords for all the children in one email (e.g., "your unique passwords: (Child1) P-XX-X-XX-B-pass1, (Child2) P-XX-X-XX-B-pass2").

If we can continue on-site recruitment for follow-up, we will use a mixed-method approach; both paper and online surveys will be available to parents for follow-up.

Depending on the response rate, UCLA paper surveys may be delivered to sites in order to increase participation. Since most sites preferred paper and the paper response rate was better for all sites, for cohort 2 follow-up and cohort 3, data collection will be conducted via paper only.

In order to expedite height and weight adipose measurements (and instrument turn around), parent consent sheets were distributed separately from parent surveys. During height and weight equipment dropoff/instrument training with preschool staff, preschool staff were instructed to ask parents to complete and return the consents on-site (prior to their child taking part in height and weight data collection), while parents were allowed to bring the parent survey home with them to complete.

Survey Reminder Emails
Cohort 1 Follow-up and Cohort 2 Baseline

#### Parent:

- UCLA Statistician compiled a list of IDs that have completed the survey/consent form as well as IDs that are in progress. UCLA Statistician sent the compiled list to the project coordinator and project assistant on Monday (previously Tuesday). Project assistant updated password tracking documents ("Year 2 Unique ID Tracker", "Year 2 - For MailChimp", "Baseline Year 2 Parent Email Tracking").
  - a. If a parent returned a completed paper survey in the previous week, and has an email on file, their email was removed from the email list.

Due to **multiple types of completion** (types following), UCLA created multiple unique reminder emails for parents to fit their completion type. Types of completion status and reminder emails following:

Families with one child:

- Parents did not complete either the survey or consent form
- Parents completed the survey but not the consent form
- Parents completed the consent form but not the survey
- Parents started the survey but did not complete the consent form

Families with multiple children at participating preschool:

- Parents completed both consent and survey for one child but did not complete either document for their second/third child
- Parents completed consent forms for all their children but did not complete the surveys for any of their children
- Parents completed surveys for all their children but did not complete the consent forms for any of their children

- 2. Once tracking documents are updated per UCLA Statistician's compiled report (#1 above), reminders are sent in the following order on Tuesday and Wednesday:
  - 1. Families with one child enrolled at the participating preschool:
    - With multiple completion types (above), email reminders were sent in the following "suborder":
      - i. Parents have not completed the survey or consent form
      - ii. Parents completed the consent form but not the survey
      - iii. Parents completed the survey but not the consent form
      - iv. Because most parents fall into one of the above 3 categories, the last group(s) that the project assistant emails are the parents that have completed any other combination of the above (e.g. [one kid]: completed consent and survey is in progress, [mult kids]: completed both documents for one child, neither document completed for other child)
  - 2. Families with two children enrolled at the participating preschool: (sub order above)
  - 3. Families with three children enrolled at the participating preschool: (sub order above)
- Once sent, the dates on which the reminders are sent are added to tracking documents.

#### Teacher reminders are sent out after all parent reminders are sent out (Wednesday/Thursday)

- 1. Same as Parent #1
- 2. Send after all Parent reminders are sent out
- Order: 1st nothing completed, 2nd- no survey, 3rd no consent, 4th- "special" (e.g., completed consent and survey in progress)

#### Parent On-site Recruitment/ Tabling Events Cohort 1 Data Collection:

Depending on the site response rate, UCLA research staff may conduct on-site parent recruitment events in order to distribute and/or collect materials during drop-off and pick-up. Since the primary outcome is BMI, we will encourage parents to complete the H&W consent on-site as well as the survey. The survey takes approximately 5-10 minutes for parents to complete (slightly longer for Spanish language surveys). It can be provided as a take-home as well. Parents would receive a gift card on the spot if they completed the survey on-site.

H&W measurements can be done during parent recruitment events, but measurements should not be shared with parents until after survey completion.

#### Pilot Testing Parent Survey Procedure

Pilot testing was conducted prior to launching the parent survey in order to obtain parent feedback and make any necessary adjustments.

All piloting materials, including procedure, can be found: Box Data Collection InstrumentsPilot Testing

## Survey Entry

Surveys are conducted on paper and entered into Qualtrics by UCLA research staff and/or interns. All paper copies are retained in the UCLA project coordinator's or project assistant's office. Due to COVID-19, electronic surveys are available and emailed directly to participants who provide an email address.

#### See APPENDIX V: How to Enter Preschool Project Data

## Unique IDs

UCLA assigns all surveys a unique ID in order to link 1) pre and post-test data and 2) parent survey data with child measurements. Unique IDs are assigned by site, by classroom/teacher, and tracked in the *Unique ID Tracker-List*.

All surveys receive a unique ID before being entered into Qualtrics and a running list of unique IDs is kept to ensure no duplication.

As surveys are received, they are immediately given a unique 7-digit ID for teacher, parents, and children and a 4-digit ID for site directors and EPAO Observations. Sites will receive a unique numeric identifier upon signing of the commitment letter, which is used to generate IDs. Participant's unique IDs are issued in the order of enrollment.

#### See APPENDIX VI: How to Generate a Unique ID

#### Unique ID Modifications due to COVID-19

#### Unique ID Modifications due to COVID-19 - Cohort 1 Follow-up and Cohort 2 Baseline

In order to protect the privacy of each electronic survey, UCLA staff will have to pre-assign an ID and password to each participant. The link and unique password will then be emailed to each participant.

A unique ID and password list will be generated by the UCLA Statistician. Once parent emails have been obtained from site, parents will be assigned an ID. All unique IDs will be tracked in a Unique ID document maintained by UCLA.

#### Unique ID Modifications starting Cohort 2 Follow-up (5/25/21):

Since most Cohort 2 sites preferred paper and the paper response rate was better for all Cohort 2 sites at baseline, beginning at Cohort 2 Follow-up (5/25/2021), data collection will be conducted via paper only. Unique IDs are assigned to participants following their enrollment.

#### Site Director Survey Entry

Site director IDs are assigned when a site enrolls in the program. Site director IDs are assigned in the order in which sites enroll. Site director IDs are used on the site director survey only. Once a site director ID is assigned, the site director survey is entered in Qualtrics. Surveys conducted on paper and entered into Qualtrics by UCLA research staff and/or interns. Data will be maintained by the UCLA statistician.

#### Cohort 1 Follow-up and Cohort 2 Baseline Survey Entry

Electronic surveys will automatically be logged into the Qualtrics system.

#### Teacher Survey Entry

Teacher IDs are assigned based on the classroom. If multiple teachers are in one classroom, lead teacher is assigned first ID for the classroom. If there are multiple teachers in one classroom but no lead teacher, teacher IDs are assigned at random. Teacher IDs are used to link pre-post data as well as link teacher survey data to teacher height and weight data. Once a teacher ID is assigned, teacher survey is entered in Qualtrics. Data will be maintained by the UCLA statistician.

#### Cohort 1 Follow-up and Cohort 2 Baseline Survey Entry

Electronic surveys will automatically be logged into the Qualtrics system.

Starting 5/25/21 (Cohort 2 Follow-up and Cohort 3), all teacher surveys were collected via paper.

#### Parent Survey Entry

Parent IDs are assigned based on their child's preschool classroom/teacher. This allows us to see if the intervention had an impact on each classroom. Parent IDs are used to link pre-post data as well as parent self-report data to child height and weight measurements. Once a parent-child unique ID is assigned, the parent survey is entered in Qualtrics. Parent ID and child are assigned a matching ID. Surveys conducted on paper and entered into Qualtrics by UCLA research staff and/or interns. Data will be maintained by the UCLA statistician.

#### Cohort 1 Follow-up and Cohort 2 Baseline Survey Entry

Electronic surveys will automatically be logged into the Qualtrics system.

## 2) EPAO and Policy Review

#### **EPAO**

EPAO citation: Ward DS, Hales D, Haverly K, Marks J, Benjamin S, Ball S, et al. An instrument to assess the obesogenic environment of childcare centers. *Am J Health Behav* 2008; 32(4): 380-6.

EPAOs should be scheduled for 1-2 weeks from In-person Meeting 1. All scheduled dates and completion dates of an EPAO logged in <u>SITE DEMOGRAPHICS AND SITE NOTES</u>. Observations take 5-6 hours each. All observations are done in teams of two. Only trained UCLA staff can conduct an EPAO. UCLA staff conducted an EPAO training August 12–14 at CPCR. <u>EPAO TRAINING</u> documents can be found on Box. All observers must complete the EPAO certification training, provided by University of North Carolina, and receive a certification score of 85% or better.

While scheduling an EPAO with the site director, UCLA research staff also send a request for policy documents. A week before a scheduled EPAO, UCLA research staff send a follow-up reminder email. Upon arrival to preschool site for an EPAO, UCLA staff requests documents again. It is ideal to have at least 3 months of menus when conducting a document review. The next steps are to collect teacher surveys and deliver parent surveys.

If a preschool has multiple preschool classrooms, the site director designates which classroom will be observed. One classroom per site; same classroom pre and post.

EPAO paperwork should be turned in to UCLA staff no later than the following business day.

University of North Carolina provided an Excel data log for entering data. They also provided the SAS programming. The main excel database has each section of the observations broken out into different tabs along the bottom. SAS combines the tabs and calculates the outcomes. Data is entered by UCLA research staff and analysis is conducted by the UCLA statistician using UNC's provided SAS code.

All EPAOs are logged on the EPAO DATA ENTRY TABLE.

#### See APPENDIX VII: EPAO

#### EPAO Modifications due to COVID-19

Due to COVID-19, the EPAO will not be conducted for cohorts 2 and 3. Policy documents will be requested after in-person meeting 1.

As of January 2022, preschools are still implementing social distancing practices and not allowing any visitors inside campus buildings. The EPAO was not included at any of the project sites due to COVID regulations.

## 3) Height and Weight Measurements

## Height and Weight Measurements

Height and Weight (H&W) measurements should be scheduled to occur within 2-4 weeks of parent survey packets delivery. H&W measurements can be conducted during parent engagement events, but measurements should not be shared with parents until after the survey has been completed.

Height is measured using a calibrated portable stadiometer. Weight is measured using a research quality calibrated digital scale. Research staff ensures calibration prior to measurement collection. Calibration is established by measuring a test subject three times on each piece of equipment to ensure all measurements are consistent across and within each piece of equipment. All height measurements are documented in INCHES to the nearest 1/8 inch and weight measurements are documented in POUNDS. Additionally, we collect each child's gender and birth date while collecting the measurements.

As students return H&W consents, a running list of who can be measured (identified by name and unique ID) is created: The *HEIGHT AND WEIGHT IDENTIFIER* (word doc) (only used at baseline cohort 1; see COVID-19 Modifications).

Identifier doc links participant name to unique ID. Unique ID is entered on the <u>HEIGHT AND WEIGHT DATA COLLECTION</u>

<u>SHEET</u> to keep documented measurements anonymous. Only students who have returned a consent form are able to participate in H&W.

See *Gift Cards* section for height and weight distribution envelopes, which are given to the teacher to give to the parents of children who participated that day. A follow-up measurement collection is scheduled for the children that were absent that day. Data are entered into *HEIGHT AND WEIGHT DATA ENTRY*.

#### See APPENDIX VIII: Height and Weight Materials

Height and Weight Modifications due to COVID-19

Height and Weight Modifications due to COVID-19 - March 2020 – September 2021, Cohort 1 Follow-up through Cohort 2 follow-up

Due to COVID-19, if UCLA staff is not allowed onto preschool property, preschool directors and teachers will be asked to conduct the measurements. A scale and stadiometer will be delivered to the preschool by UCLA staff. A training PowerPoint has been put together to train the preschool staff. The PowerPoint can be sent ahead of time to a site and must be reviewed with whomever will be conducting the measurements during equipment drop-off. A link to complete a 5-question comprehension check is provided at the end of the PowerPoint. All staff collecting the measurements will be asked to review the training. A list of the students who have consented will be provided to the site in order to collect data. The participant name's will be provided, rather than the unique ID, for ease of data collection for the site director. Data will be logged by Unique ID in the Data entry excel spreadsheet.

In order to expedite height and weight adipose measurements (and instrument turn around), parent consent sheets were distributed separately from parent surveys. During height and weight equipment dropoff/instrument training with preschool staff, preschool staff were instructed to ask parents to complete and return the consents on-site (prior to their child taking part in height/weight data collection). Parents were allowed to bring the parent survey home with them to complete.

Scales and stadiometers were calibrated to assess validity.

Height and Weight Modifications - UCLA field research restrictions lifted September 2021, Cohort 3 baseline

UCLA's restrictions for field research activities were lifted in the Fall of 2021, allowing the project to return to the originally planned approach of having UCLA staff members conduct the height and weight measurements. All UCLA staff members are fully vaccinated against COVID-19 and complete a daily symptom monitoring survey prior to entering UCLA campus and any participating study sites. Participating sites that had on-going height and weight consent collection prior to the lifted restrictions, were notified of the lifted field restrictions via phone. UCLA research staff followed a script (hyperlinked script: "Preschool Cohort 3 Height weight measurements by UCLA staff FINAL 9 30 21".) to notify sites

If a participating site has policies against off-campus visitors, preschool directors and teachers will be asked to conduct the measurements following the above COVID-19 modifications. If this approach is used, UCLA staff members will observe the measurements either in person, via Zoom, or another video conferencing program in order to provide any necessary guidance to the teachers as they conduct the measurements.

#### See APPENDIX IX: SCALE CALIBRATION PROTOCOL

#### Gift Cards

All gift cards must be documented before distributed in <u>GIFT CARD TRACKING</u>. The gift card 15-digit serial number is documented, and a corresponding shorthand number is assigned.

Once participant surveys have been received by UCLA, gift cards will be distributed to the preschool. Gift cards are placed in an envelope along with a thank you note, sealed, and labeled with the site, parent name, and child's name.

Prior to delivering gift cards to sites, UCLA staff prepare a gift card sign-out sheet (*GIFT CARD LOG*). The gift card sign-out sheet is prefilled out by UCLA staff with the participant's name and pre-assigned gift card number. Two copies of the sign-out log are delivered to the site (one for the director to sign as proof of delivery from UCLA, and the second to leave with the director to have participants sign for their gift card). All participants must sign for a gift card next to the corresponding number on their card.

#### **Gift Card Amounts**

| For: | Pre Amount: | Post Amount: |
|---------------------------|-------------|--------------|
| Parent survey | \$10 | \$20 |
| Child height and weight | \$5 | \$5 |
| Teacher survey | \$10 | \$25 |
| Teacher height and weight | \$5 | \$5 |
| Site Director survey | \$10 | \$25 |

## Phase III: Randomization and Implementation

### Randomization of Sites

Randomization will occur once most sites have completed the EPAO and the NAPSACC surveys. Sites are stratified by the following: CACFP (aka food program) participation, number of site provided meals, and preschool size.

Regardless of randomization, all sites will participate in pre/baseline (at beginning of the school year) and post/follow-up (at the end of the school year) data collection activities, including:

- 1) Site Director/ NAPSACC survey
- 2) Teacher surveys
- 3) Parent surveys
- 4) Height and Weight Measurements
- 5) EPAO and Policy Review (Cohorts 2 and 3 only Policy Review due to COVID)

<u>Sites that are randomized to the intervention arm</u> will receive materials at the beginning of the school year. Materials include:

- 1) Intervention materials (Sesame Street binder and parent materials)
- 2) Program banner
- 3) 2-liter pump hand sanitizer (with ABC Healthy Me Sticker)
- 4) Coaching (1-2 times a month per teacher per site for up to an hour)
- 5) Stipend and supply allotment

<u>Sites that are randomized to the delayed-intervention arm</u> will receive materials at the end of the school year. Materials include:

- 1) Intervention materials (Sesame Street binder and parent materials)
- 2) Stipend and supply allotment
- 3) Abridged coaching (1-2 sessions at the end of the school year)
  - a. Cohort 2 sites that were randomized to the delayed-intervention arm are to receive abridged coaching throughout the following school year. (1 session every other month throughout the school year). This group will receive coaching through our "cohort coaching model"; sites will receive coaching in the same

sessions as other sites in order to promote support between schools during the months they will not receive nutrition and physical activity coaching.

### **Implementation**

Implementation is guided by the A-B-C Healthy Me Required and Supplemental Component Table and the RE-AIM table.

- A-B-C HEALTHY ME REQUIRED AND SUPPLEMENTAL COMPONENT TABLE
- RE AIM TABLE

\*Since this is an implementation science project, the goal of this implementation is to apply a gentle touch in guiding sites to make permanent, sustainable change.

Implementation begins with an initial coaching session to introduce the program to teachers and discuss the curriculum. The coach works with the site director to establish if the first coaching session occurs with the site director and the teachers together or separately. At least one coaching session occurs with the site director to address the supplemental components of interest and address policy changes to be made. During the initial coaching session, the site staff and the coach review the Component Table and select targeted activities.

#### Implementation focuses on:

- Improving health policies per the A-B-C COMPONENT TABLE
- Integration of SESAME STREET HEALTH HABITS FOR LIFE into curriculum
- Teacher modeling of healthy behaviors
- Parent engagement via events and monthly handouts
  - o **PARENT ENGAGEMENT TRACKER**
  - **O PARENT MONTHLY HANDOUTS**
  - PARENT MONTHLY BOOKLETS

#### Implementation Tracking

#### Implementation monitored and documented via:

- <u>COACHING SITE SUMMARY</u>: meant for the coach to document the subject matter of the coaching session, the action plan to attain goals, and next steps. Multiple subject matters may be discussed during one coaching session. Subject matters include: curriculum and learning activities, resources, family engagement, education or professional development, policy, practice, and environment.
  - The coach completes this with whomever is receiving the coaching, which is most often the teachers.
  - o The coach will enter the data into SurveyMonkey, which is managed by CCRC.
- **QIP FORM(S)**: the quality improvement plan. This is the plan the teacher will use to implement what they learned in coaching and how they will achieve the plan goal.
  - The coach completes this with whomever is receiving the coaching, which is most often the teachers.
  - The coach will enter the data into SurveyMonkey, which is managed by CCRC.
- <u>TEACHER TRACKER</u>: a weekly report of activities the teacher conducted in the classroom. Planned
  activities are captured and submitted on the lesson plan. This will allow us to know the fidelity of
  implementation.
  - o The teacher fills this out and submits weekly via email or google doc, per site preference.
  - UCLA will enter the data into the <u>COACHING DATA TRACKER</u>
- <u>LESSON PLANS</u>: allows teachers to plan for how to integrate Sesame Street into their planned activities. Teachers will work with the coach to identify which lessons and where in their existing schedule they can integrate these activities.

- The teacher fills out either on their own or with the coach at first. The teacher submits via email weekly (preferred, but site dependent).
- o Lesson plans will be scanned and uploaded to Box.
- <u>COACHING VISIT TRACKER</u>: allows the coach to track how many visits they have had with each teacher from each site.
- **PROGRESS NOTES**: kept to maintain notes of what is going on at each site.

## Coaching

The coach will ideally meet with each teacher at a site, twice monthly, for one hour each visit, depending on availability. The coaching happens on a strength base approach and meeting the teacher where he/she is. Building a relationship is part of the coaching as it helps teachers feel supported and connected. The initial coaching visit is about the coach and the teacher establishing a connection and talking about classroom routines and program structure. Logistics about what coaching sessions will look like is also discussed with the teacher.

Coaching has a few moving parts. There are goals that are created by the teacher with the support of the coach. These goals are specific, measurable, attainable, relevant and time bound. The goals are also developed based on the requirements of the program and the need of the classroom from the coach's observation. These goals are developed and tracked on our Quality Improvement Plan (QIP) as well as every follow up for that goal. Depending on the goals, a teacher may be working on more than one goal at one given time, considering that some goals will have a very short timeline.

After every visit the coach completes a site summary visit where data on the one-hour visit is completed; this data consists of duration of the visit, the number of adults in the classroom during the visit as well as the number of children in attendance during the visit, if children are present. The coach also connects with the center director after each coaching session with teachers to keep the director informed of all of the coaching activities, teacher goals and provides resources and coaching in the administrative aspect of the program.

Once the control sites have completed their site director and teacher surveys, they will be contacted for coaching. Coaching will be abridged, approximately two 1-hour sessions, to help teachers get an understanding of the Sesame Street curriculum and how to implement it themselves as well as meeting with each site director to discuss policy recommendations.

#### Coaching Modifications due to COVID-19

#### Coaching Modifications due to COVID-19- March 2020 – present (January 2022)

Coaching has currently shifted to accommodate the current situation with the COVID-19 pandemic, being sheltered in place and not being able to conduct visits. Coaching is now being done virtually and over the phone and it looks a little different. Teachers are experiencing uncertainty, anxiety and stress, most of the coaching conversations begin with the coach listening and offering support in any way possible. We are currently working to develop a different approach to engage not only teachers but also the families. As of January 2022, coaching for cohort 3 is still conducted virtually.

All Teacher materials were moved to a website: abchealthymeteacher.wordpress.com

#### Coaching Modifications for Cohort 2

Cohort 1 control sites are being given the opportunity to enroll for a second year as an intervention site. Their follow-up data from their first year will act as baseline data for their second year. Once control sites have started their data collection and are scheduling their height and weight measurements, they will be contacted for coaching. If a site does not participate in follow-up data collection, they will not be allowed to receive coaching.

Additionally, control sites will be provided Health and Safety Coaching. In general, the coach could possibly facilitate training addressing some of the most common deficiencies found by Community Care Licensing and by the

most common trends amongst providers found by the coach during visits. This would help support and enhance Health and Safety practices on a daily basis by doing the following:

- Conduct Health and Safety screenings
- Identify areas of focus based on the needs of the site and implement corrective action plans
- Support in implementing Community Care Licensing Title 22, best practices and Caring for Our Children National Health and Safety Performance Standards as well as new regulations and compliance with Health and state post COVID 19
- Collaborate with provider/teachers and program coach to ensure high quality operation of program based on findings and recommendations
- Provide resources to support the implementation of Health and Safety practices
- Support providers/teachers with any updates made by Community Care Licensing, Centers for Disease Control and Department of Public Health
- Maintain communication with provider and program coach to ensure compliance

### Family Child Care (FCC) Coaching – Cohort 2

FCC coaching will be scheduled as a group, bringing together FCCs to collaborate as a cohort. Cohort sessions will begin after the first individual coaching visit with each site and occur monthly. Coaching visits with individual providers will happen based on the need of the provider and the discretion of the coach if she feels providers need additional support.

Goals addressing the need and requirement of the program will be created in order to conduct the cohort coaching (all providers will be coached on implementing the same goals at the same time). The strategy behind the cohort coaching is to be able to conduct visits with providers as a group so that they may also be of support to each other throughout the program year.

#### Coaching Data Entry

Data collected from coaching forms (site summary and QIP) is entered into SurveyMonkey and run by CCRC. The teacher tracker and lesson plans are submitted weekly by the teacher to the coach and scanned and uploaded to Box. A tracking system allows the coach to know which sites have turned in their lesson and plans and trackers.

## Parent Engagement

As part of the program, sites are required to host two parent engagements each school year. Parent engagement events are meant to bring preschool parents together to engage in a physical activity or nutrition learning. Depending on the site, each classroom may hold a parent engagement event for the parents of that classroom or the whole school may host for all parents. Events may include: Zumba, yoga, dance cardio, healthy snacks, rethink your drink, etc.

#### Parent Engagement Modifications due to COVID-19

Starting May 2020: Due to COVID-19, parent engagement events are available via Zoom.

Starting March 2021, Cohort 2 sites conducted parent engagement events in-person, online, or as a "takehome" option in accordance with their school's social distancing policies. Coaches work with the site directors to schedule events, send event flyers, and notify parents. CCRC coaches lead these events. CCRC may also reach out to outside contractors who may be willing to lead an event.

#### Parent Website

The A-B-C Healthy Me website (<a href="www.abchealthyme.wordpress.com">www.abchealthyme.wordpress.com</a>) provides our intervention sites with resources they can share with parents and parents can come back to for relevant health information. The information available on the website has been created by the A-B-C Healthy Me team and/or was recommended for use by the CCRC coaching team. Links to external resources are provided throughout the website so parents can choose which content to

use. Resources and links can be updated by UCLA at any time to provide our participants with up-to-date health information.

The main pages of the website include: Nutrition Resources; Physical Activity Resources; downloadable versions of all the A-B-C Healthy Me Parent Booklets (in English and Spanish); and at-home learning resources. Additionally, there is a COVID-19 page with links to helpful family COVID-19 resources including the Center for Health Equity resource page and the CA Department of Health COVID website.

The A-B-C Healthy Me website will be made available to parents through their preschool site. Sites selected for intervention will be provided with the URL to share with parents. It will also be included in all A-B-C Healthy Me resources sent to parents. Parents can then access resources, find helpful information, and download parent booklets.

We have selected to launch the website in "hidden" mode so that the URL will not be searchable or available on major search engines (such as Google or Yahoo). In order to limit barriers to access, password protections will not be required for participants to gain access to this website. We do not expect participants to share this information outside of their school and we will discuss limiting sharing of this resource with the site director during the coaching meeting.

## Phase IV: Follow-up Data Collection

## Follow-Up Data Collection

Follow-up data collection will begin with control sites and then rollout at intervention sites. This will allow us to efficiently collect follow-up data at each site while allowing the intervention to continue with as much time as possible.

#### Cohort 1 Follow-up Data Collection Modifications due to COVID-19

Due to COVID-19, in-person cohort 1 follow-up data collection paused, leaving surveys to be distributed electronically. In order to protect the privacy of each electronic survey, UCLA will have to pre-assign an ID and password to each participant. The link and unique password will then be emailed to each participant. Paper surveys can be delivered to sites that do not communicate via email with parents or do not believe their parents will participate electronically.

#### Cohort 2 Data Collection Modifications due to COVID-19

Cohort 2 baseline data collection initially was collected electronically. However, many sites requested that paper surveys also be distributed to their parents and teachers. Most Cohort 2 sites preferred paper and the paper response rate was better for all Cohort 2 sites at baseline. Beginning at Cohort 2 Follow-up data collection (5/25/2021), will be conducted via paper only. Unique IDs are assigned to participants following their enrollment

Additionally, parents that did not participate in baseline data collection activities will be eligible to participate in follow-up activities. Many sites saw great turn over in children during the start of the pandemic, leaving many of the baseline participants to no longer be enrolled at the site for follow-up. However, new parents have enrolled and thus may still be able to provide insights into the preschool environment.

## Follow-up Surveys

#### Paper Follow-up Surveys

All surveys will be delivered at the same time to a site (parent, teacher, and site director). Teacher and site director surveys will be collected one week after delivery. Parent surveys will also begin collection one week after delivery and last for 2-3 weeks with a weekly pick up from the site director. Parents who did not participate in the baseline survey may still participate in the follow-up survey.

Starting 5/25/21 (cohort 2 follow-up and cohort 3), data collection will be conducted via paper only.

#### Electronic Follow-Up Surveys- Cohort 1 Follow-up

In the event we are unable to distribute surveys directly to participants on-site (i.e., COVID-19), we will ask site directors if they are able to circulate surveys through their parent contact network (i.e., Email, app-based, etc.) and to their teachers. For parents who provided their contact information at enrollment, we will directly send their survey link to them via email. The email will contain the link to the survey as well as required password to enter the survey. The link and password will be assigned to their unique ID.

Otherwise, other parent emails must be collected from the site in order to provide parents with the survey link and unique password. A *PARENT or TEACHER EMAIL COLLECTION FLYER* will be emailed to the site director to email to their parents. The flyer provides information on the program and explains the opt-out model of email collection. If a parent does not want to participate, they are told to let their site director know. After a week, UCLA will reach out to collect parent emails from the site director.

Once parent emails have been collected, UCLA will send each parent the <u>PARENT BASELINE SURVEY LINK AND</u>

<u>PASSWORD EMAIL</u> explaining the program and providing the survey link and password. Email addresses and unique survey information will be extracted from our Unique ID tracking data and compiled using a Python code. Emails will be sent to participating parents via the webhost, MailChimp, and will contain the link to the survey as well as the required password to enter the survey. The link and password will be assigned to their unique ID.

If we are able to continue on-site recruitment for follow-up, we will use a mixed-method approach; both paper and online surveys will be available to parents, teachers, and directors for follow-up.

Beginning 5/25/21, cohort 2 follow-up and cohort 3 data collection will be conducted via paper only.

## Follow-up EPAO

Control EPAOs will occur at the beginning of the month and intervention site EPAOs will be conducted at the end of the month. Ideally, the same team that conducted the baseline EPAO will conduct the follow-up EPAO. Follow-up EPAOs for intervention sites may be conducted while coaching activities are still on-going; however, control sites follow-up EPAO must be conducted before contact with coaching.

In the event the follow-up EPAO cannot be conducted in the same "school year" as the baseline (i.e., COVID-19), follow-up EPAOs will be conducted as soon as possible. Ideally, the same teacher will be observed at both the baseline and follow-up. If the same teacher is unavailable, another preschool teacher will be selected by the site director for observation.

## Follow-up Height and Weight

Follow-up height and weight measurements will follow the same protocol as baseline measurements. Multiple sessions may occur at each site in order to collect all children's measurements. Participants who did not participate in baseline measurements may still participate in follow-up measurements. UCLA research staff will distribute consent forms on-site at measurements.

In the event the follow-up height and weight measurements cannot be conducted in the same "school year" as the baseline (i.e., COVID-19), follow-up height and weight measurements will be conducted as soon as possible. Children who participated in baseline may still be on-site but in a different classroom. Additionally, new participants will be recruited to participate in the follow-up measurements.

## **Phase V: Evaluation**

### **Program Evaluation**

Program evaluation will be assessed periodically during the intervention period and will be guided by the **RE-AIM table** 

#### **Process Evaluation**

#### Implementation monitored and documented via:

#### • COACHING SITE SUMMARY

- This summary is meant for coaches to document the subject matter of the coaching session, the action plan to attain goals, and next steps. Multiple subject matters may be discussed during one coaching session. Subject matters include: curriculum and learning activities, resources, family engagement, education or professional development, policy, practice, and environment.
- The coach completes this with whomever is receiving the coaching, most often the teachers.
- The coach will enter data into SurveyMonkey, managed by CCRC.

#### • QIP FORM

- This form is the quality improvement plan. This is the plan the teacher will use to implement what they learned in coaching and how they will achieve planned goals.
- o The coach completes this with whomever is receiving the coaching, most often the teachers.
- o The coach will enter data into SurveyMonkey, managed by CCRC.

#### • TEACHER TRACKER

- This is a weekly report of what activities the teacher conducted in the classroom. Planned
  activities are captured and submitted in the lesson plan. This will allow us to know the fidelity of
  implementation.
- The teacher fills this out and submits weekly via email or google doc, per site. preference.

#### • LESSON PLAN DOCUMENTS

- These documents allow the teacher to figure out how to integrate Sesame Street into their planned activities. Teachers will work with the coach to identify which lessons and where in their existing schedule they can integrate these activities.
- The teacher fills out either on their own or with the coach at first. The teacher then submits via email weekly (preferred, but site dependent).

#### Outcome Evaluation

Program outcomes include the following:

#### Effectiveness:

- Primary: Change in zBMI of preschool students
- Secondary:
  - Change in preschool student nutrition as reported by parents
  - Change in preschool student physical activity as reported by parents
  - Change in zBMI of preschool teachers
  - Change in preschool teacher nutrition
  - Change in preschool teacher physical activity

#### Implementation:

- Primary: EPAO scores (discontinued due to COVID)
- Secondary: NAP SACC scores

## APPENDIX I: Initial Director Call Talking Points

#### The initial call entails:

- Explaining the partnership between UCLA and CCRC
- □ Reviewing program goals and expectations
  - o Program goals are meant to be flexible to the needs of each site
- Clearly explaining that <u>sites will be randomized</u> into two arms (intervention and delayed intervention)
  - o All sites will eventually receive the intervention and stipend.
  - Sites that are randomized into the delayed-intervention group will complete surveys, height and weight measurements, and observations at the beginning and end of the year; however, they will not receive program materials or stipends until the end of the school year. This also means these sites will receive abridged coaching.
- Assessing readiness to agree to participation
- □ Referring to "Why Should a Site Participate?" section below for additional information
  - Sites that do not agree to participation during the initial call will receive a follow-up call a week later to gauge interest.
  - o Encourage site directors who are unsure to discuss with their teachers

#### Why Should a Site Participate?

- Sites will set own nutrition and physical activity goals
- Sesame Street Healthy Habits for Life is a nationally recommended and evidence-based curriculum
- Sites will receive support throughout the duration of the intervention as well as \$500 to purchase supplies/resources to support the implementation of nutrition and physical activity policies
- Trusted CCRC coaches will assist with curriculum/lesson planning to support classroom learning
- Childhood obesity can affect development, brain function, self-esteem, and increase disease risk
- Childhood nutrition and physical activity preferences are typically established during preschool years and track into adulthood, leaving children who become overweight/obese to be at a fivefold increased risk of being overweight/obese adults<sup>2</sup>
- 20% of preschool aged children in Los Angeles County are overweight or obese<sup>1</sup>
- Nearly 61% of children under the age of 5 in the U.S. are enrolled in nonrelative, center-based care where they spend an average of 33 hours per week and receive majority (2/3) of meals<sup>2</sup>
- CACFP new recommendations (effective as of Oct. 1, 2017) include<sup>3</sup>:
  - o Both fruits and vegetables (or two different vegetables) served at lunch
  - o Juice may be served and counted as fruit component of the meal, but is limited to once per day
  - o One serving of whole grain-rich grains must be served each day
  - o Grain-based desserts, such as cookies, cakes, pies, are no longer reimbursable as a grain
  - Meal patterns limit added sugar by requiring unflavored milk only for children 0-5 and limiting sugar in readyto-eat cereals and yogurt
- Staff modeling (specifically sitting with children and eating the same food as children) associated with higher vegetable and fruit intake<sup>2</sup>

#### APPENDIX II: Initial Call

#### When reaching out to a site to set up an initial call:

- 1. Copy and paste the **site recruitment script** in the body of an email and attach the **site recruitment flyer** to the email and send to the site director before the initial call.
  - SITE RECRUITMENT SCRIPT
  - SITE RECRUITMENT FLYER

#### **During the initial call:**

- 1. Complete the <u>INITIAL RECRUITMENT CALL COLLECTION</u>. This needs to be filled out during each call to a site.
  - Have the site recruitment script and flyer available to review. (<u>SITE RECRUITMENT SCRIPT</u> and <u>SITE RECRUITMENT FLYER</u> on Box)
- 2. Schedule in-person meeting 1

#### After Initial call (within 24 hours),

- 1. Initial call data logged in the INITIAL CALL/RECRUITMENT DATA LOG
- 2. Send email containing:
  - Calendar invite for in-person meeting 1
  - Copy and paste:
    - SITE AGREEMENT SCRIPT
    - **O SITE DIRECTOR PARTICIPATION LETTER**
    - TEACHER PARTICIPATION LETTER\*

<sup>\*</sup>The site director will forward to teachers and paper copies are also brought to in-person meeting 1

## APPENDIX III: In-Person Meeting 1

#### **Cohort 1: At In-Person Meeting 1:**

- 1. Bring **Teacher Sample Binder** and **Site Folder** containing:
  - At least 3 copies of the <u>TEACHER RECRUITMENT LETTER</u> (remember to add the name of the school and date)
  - SITE COMMITMENT LETTER
  - ACTIVITY TABLE
  - SITE DEMOGRAPHICS PAPERWORK
  - SITE DATA COLLECTION PROCESS FORM
- 2. Deliver:
  - Site director Survey Packet:
  - Teacher Survey Packet:
    - i. Teacher participation letter
  - \*Document date of delivery in INITIAL CALL/RECRUITMENT DATA LOG
- 3. Complete:
  - Schedule EPAO observation day for within two weeks of in-person meeting 1
  - SITE COMMITMENT LETTER
  - SITE DEMOGRAPHICS PAPERWORK
  - SITE DATA COLLECTION PROCESS

Site Demographics and Data Collection form logged in Site Demographics and Site Notes

#### **Cohort 2: At In-person Meeting 1:**

#### RECRUITMENT POWERPOINT

#### After in-person meeting 1, email (link script) site directors:

- 1. Calendar invite for data collection meeting
- 2. Site director and teacher participation letters
- 3. Participation agreement
- 4. List of documents to submit

## APPENDIX IV: Participant Survey Packets

- Site director Survey Packet:
  - i. SITE DIRECTOR PARTICIPATION LETTER
  - ii. SITE DIRECTOR SURVEY CONSENT
  - iii. NAPSACC SURVEY
- Teacher Survey Packet:
  - i. TEACHER PARTICIPATION LETTER
  - ii. TEACHER SURVEY CONSENT
  - iii. TEACHER H&W CONSENT
  - iv. TEACHER SURVEY (\*Remember to add name of school and date)

#### PARENTS:

\*Parent materials for print and a sample envelope can be found in the top cabinet of the filing cabinet at the back of A2-125E

- o ENGLISH
- o SPANISH
  - PARENT PARTICIPATION LETTER
    - Print in color on white paper
  - PARENT INFORMATION SHEET
    - Print on white paper
  - PARENT SURVEY
    - Print on green paper
  - CHILD HEIGHT AND WEIGHT CONSENT
    - Print on blue paper
  - CONTACT SHEET
    - Print on yellow paper

<sup>\*</sup>Put "PARENT SURVEY ENVELOPE LABELS" label and "EARN \$25 IN GIFT CARDS. LOOK INSIDE." sticker on front of each parent survey packet

## APPENDIX V: How to Enter Preschool Project Data

There are 3 surveys for each preschool project site:

- 1. Site Director (NAPSACC)
- 2. Teacher
- 3. Parent

#### When entering surveys:

- Enter all data AS IS (to the best of your ability).
- When entering survey ID, include dashes.
- If two answers are selected, default to the right most answer. Definition of "right most answer" following:
  - o If answer choices available are: □ agree □neither agree nor disagree □ disagree
    And participant checks two boxes (e.g.: □ agree ☑ neither agree nor disagree ☑ disagree), key the right most answer: "disagree"
- If **two answers are selected but are opposing** (i.e., agree and disagree) or have a gap between them in answer choices, key the average and put a note in the notes section.
  - Ex. If someone keys both 'Never' and 'Sometimes', average to 'Rarely'
  - Ex. If someone keys both 'Agree' and 'Disagree', average to 'Neither agree nor disagree'
- If an answer is blank, key 'refused to answer' unless otherwise specified
- If a **range is written** in (i.e., 60-90 minutes), feel free to key the average (75) but note the range in the notes section as such: ex. = #9: 60-90
- Refused to answer vs. don't know
  - Refused to answer (99):
    - If something is blank or missing, but all other data in the section has been filled out
    - If something is blank or missing because it is sensitive information a participant might not want to share with us
  - Don't know (88):
    - If something is blank or missing because it might not be available information to the participant (i.e., height and weight).
- ALWAYS initial and date a survey after completion.
- Please **do not abandon** a survey in the middle of entry.
- If entering SPANISH surveys, enter all notes in Spanish. They will be translated on the back end.
  - During Cohort 2 follow-up data collection, project team transitioned to translating notes before entering data in order to expedite analysis at a later date.
- When entering multiple teacher or site director surveys, fully close internet browser (including all open windows) to reset the link.
- If **height** has a fraction,  $\frac{1}{2}$  or > = round up; less than  $\frac{1}{2}$ , round down.
- If only feet for height is entered and inches is left blank, assume it is a whole number. Do not put refused to answer (99) for inches.
- If parent enters child's age as parent's age, mark as refused to answer (99) and write a note.

#### **How to Write a Note:**

- Please keep notes to no more than 92 characters.
- We need to know exactly how the question was answered; we will know what you inputted because we will see it in the data report.
  - Here is an example:
    - Instead of keying this (256 characters).

      For #11, participant answered 60+, I inputted 60. For #12, participant answered 3+, I inputted 3.

      For #13, participant answered 1+, I inputted 1. For #14, participant answered 7+, I inputted 7.

      For #15 weight, participant put in parenthesis (I'm pregnant)

- Use this (63 characters).
   #11: 60+, #12: 3+, #13: 1+, #14: 7+, #15weight: (I'm pregnant)
- Abbreviations:
  - Hour = hr
  - Week = wk
  - O Minute = min
  - O Month = mon
  - Never = nvr
  - Several Times per month = svrl x/ mon
  - Several Times per week = svrl x/ wk
  - Every day = evry day
  - More than once a day = > 1/ day
  - Disagree = dagr
  - Somewhat disagree = swdagr
  - Neither agree nor disagree = nor
  - Somewhat agree = swagr
  - Agree = agr
    - Ex. Abbreviation note: #5: swdagr & swagr

#### EPAO:

- If variable is numeric and answer is blank, no, or N/A, enter 0.
- If variable is character and answer is blank, missing, or NA, enter space space (or enter space (x2).
- If outdoor time was cancelled due to fire related atmosphere, mark the reason as "It was too hot"
- EPAO\_C14\_1t5\_J on excel sheet should be space space (or two spaces)
  - o It says EPAO\_C14\_1t5\_I on the data dictionary, which should be a character variable
- Decimals are OK

## APPENDIX VI: How to Generate a Unique ID

#### Format for site director and EPAO observations: X-XX-X

- 1. Digit 1: Participant type:
  - D = Site Director
  - E = Observation/EPAO
- 2. Digit 2-3: Site ID (01-99)
  - a. Schools assigned ID at In-person meeting 1
- 3. Digit 4: Pre/Post A = Pre; B = Post

For site directors: pre-post survey

For observation: pre/post EPAO

Ex. E-01-A = Observation, Site 1, pre-implementation survey

Ex. D-02-B = Site Director, Site 2, post-survey

#### Format for survey: X-XX-X-XX-X

- 1. Digit 1: Participant type:
  - T = Teacher
  - P = Parent
  - C = Child
- 2. Digit 2-3: Site ID (01-99)
  - a. Schools assigned ID at In-person meeting 1
- 3. Digit 4: Participant Classroom (1-9)
  - a. Classrooms assigned number at site enrollment
- 4. Digit 5-6: Participant # (01-99)
- 5. Digit 7: Pre/Post A = Pre; B = Post, C = Post-Follow-up Only (participant recruited at follow-up, did not participate in baseline data collection (examples for post-IDs ending in C below)

For teachers and parents: pre-post survey

For children: pre/post height and weight measurement

Ex. <u>T-01-1-03-A</u> = Teacher, Site 1, Classroom 1, Teacher 3, <u>Pre-survey</u>

Ex. <u>T-06-1-02-A</u> = Teacher, Site 6, Classroom 1, Teacher 2, <u>Pre-survey</u>

Ex. <u>P-**01**-2-11-B</u> = Parent, **Site 1**, Classroom 2, <u>Parent 11</u>, <u>Post-survey</u>

Ex. <u>C-01-2-11-B</u> = Child, Site 1, Classroom 2, Child 11, <u>Post-survey</u>

Post ID ending in C:

If a participant is newly recruited at follow-up (no baseline participation), their follow-up ID will end in -C rather than ending in -B. ID format follows the above convention for linking participant to site number and classroom.

Ex. If we receive a consent form, a survey, and/or height weight measurements for a participant at baseline, their Follow-up ID will end in -B. If we do not receive any materials or data on a participant, their follow-up ID will end in a -C.

Example: ID assignment follows above convention to link participant to site and classroom

| | X = reco | eived, blank | = not received | | _ |
|---|---|---|---|---|---|
| Baseline<br>Unique ID | Baseline<br>survey | Consent | Baseline ht/wt measured | Follow-up<br>Unique ID | |
| T-01-1-03-A | Х | Х | Х | T-01-1-03-B | All materials/data received at baseline = follow-up ID ending in B |
| T-06-1-02-A | | Х | X | T-06-1-02-B | Consent + ht/wt measured at baseline = follow-up ID ending in B |
| T-07-5-01-A | Х | | | T-07-5-01-B | Survey received at baseline = follow-up ID ending in B |
| C-07-6-02-A | | Х | | C-07-6-02-B | Consent received at baseline = follow-up ID ending in B |
| C-01-2-11-A | | | | C-01-2-11 <b>-C</b> | No baseline data/participation = follow-<br>up ID ending in C |

## APPENDIX VII: EPAO

#### At EPAO:

- 1) Collect site director and teacher surveys.
  - a. Deliver site director and teacher **GIFT CARD LOG**
- 2) Conduct EPAO:
  - a. Each observer must have an EPAO binder containing:
    - EPAO OBSERVATION PACKET
    - EPAO DOCUMENT REVIEW PACKET
    - EPAO TABLE OF CONTENTS
    - EPAO REFERENCE DOCUMENT
    - <u>EPAO PROTOCOL AND PROCED</u>URE
    - EPAO INFO SHEET
- 3) Deliver Parent Survey Packets

## APPENDIX VIII: Height and Weight Materials

When conducting H&W measurements at sites, make sure to have the following:

- o <u>HEIGHT AND WEIGHT IDENTIFIER</u>
- o <u>HEIGHT AND WEIGHT DATA COLLECTION</u>
- o HEIGHT AND WEIGHT PROCEDURE DOCUMENT
- o <u>HEIGHT AND WEIGHT PROVIDER TRAINING</u>
- o HEIGHT AND WEIGHT ACTIVITY SHEET
- Weight scale
- o Stadiometers
- o At least 2 pens
- o Envelopes with gift cards and gift card log
- o Equipment disinfectant
- o Extra height and weight consent forms

# APPENDIX IX: Scale Calibration Summary Scale Summary – 5/13/21

- Cohort 1 baseline:
  - o CPCR had three scales at the start of the project.
    - Scales came research calibrated.
    - Internal weight comparison across the three scales yielded same outcome weight across all three scales.
    - Only UCLA research staff handled the scales. UCLA research staff conducted onsite measurements for all Cohort 1 baseline height and weight measurements.
- Cohort 1 follow-up/Cohort 2 baseline:
  - o COVID-19 change:
    - UCLA research staff decided to leave scale at sites for preschool staff to collect measurements given the COVID-19 social distancing protocols.
      - Scales were numbered and labeled following the decision to leave scales at sites to adhere to social distancing protocols.
      - UCLA staff delivered scales to participating sites and trained the preschool staff following the project's anthropometric data collection procedures.
    - UCLA research staff purchased 3 additional Detecto 550 scales.
      - Detecto accidentally sent 6 scales in shipment (the 3 DR550C that we ordered and 3 additional DR400C. DR400Cs were stored at CPCR and not deployed into the field).
- Total of 9 scales as of 5/12/21 present:
  - 1. Detecto DR550C (n = 5) = scales 1-3, 5, and 6
  - 2. Tanita BWB-800 (n=1) = scale 4
  - 3. Detecto DR400C (n = 3) = scales 7-9
  - Scales #1-5 were stored in the office between 02/19/2020 10/07/2020 and 02/26/2021 present.
  - Scale #6 was stored in the office between 02/19/2020 10/07/2020 and has been with a UCLA staff member for delivery from 01/26/2021 – 5/13/2021.
  - Scales #7-9 have not been in the field and have remained in storage at CPCR.
     As of September 2021- present: (Beginning of cohort 3 baseline height and weight data collection), scales #7-9 were used in the field

#### Scale Calibration Summary

- Cohort 1 baseline/Cohort 1 follow-up/Cohort 2 baseline:
  - Before scales were deployed in the field, an internal weight comparison across the research calibrated scales was conducted by the Project Coordinator and Project Assistant using own body weight. All scales yielded the same outcome weight.
- Cohort 2 follow-up/Cohort 3 baseline:
  - O5/04/2021 05/06/2021: During Cohort 2 Follow-up preparation, scales #1-5, #7-9 were assessed for reliability within each scale and between scales. Following the project's data collection procedure, two UCLA staff members weighed themselves three times on each scale, allowing the scale to zero out between measurements. Staff members repeated this procedure over 3 days to assess instrument drift. This assessment yielded consistent readings within each of the scales 1-5, 7,8 and between these 7 scales. Scale #9 consistently read staff members' weight around 2 lbs. below the average reading of scales 1-5,7-8. Scale 6 was unavailable for comparison.
  - 05/10/2021: UCLA staff contacted Detecto and Tanita technical support via phone to inquire about lowering the scales' calibration limits (listed below). Technical support staff at both companies informed staff members that calibration limits cannot be adjusted to a lower threshold.

| Scale Brand and Model | Required Calibration weight (kg) | Required Calibration weight (lbs.) |
|---|---|---|
| Detecto DR400C | 120 | 440 |
| Detecto DR550C | 200 | 441 |
| Tanita BWB-800 | 200 | 440 |

• 05/11/2021: Scales assessed with 50 kg calibration weights. Assessment was repeated twice for each scale. This assessment found that scales 1-4 and 6-8 were calibrated. Scale #5 read 0.1kg below calibration weight. Scale #9 was found to be out of calibration (below). Scale #6 was with a UCLA staff member and was assessed on 5/13/21.

| Scale<br>Number | Scale Brand and model | Calibration weight | Output<br>Measurement 1 | Output<br>Measurement 2 |
|---|---|---|---|---|
| 1 | Detecto 550 | 50kg | 50 kg | 50 kg |
| 2 | Detecto 550 | 50kg | 50 kg | 50 kg |
| 3 | Detecto 550 | 50kg | 50 kg | 50 kg |
| 4 | Tanita BWB 800 | 50kg | 50 kg | 50 kg |
| 5 | Detecto 550 | 50kg | 49.9 kg | 49.9 kg |
| 6 | Detecto 550 | 50kg | 50kg | 50kg |
| 7* | Detecto 400 | 50kg | 50 kg | 50 kg |
| 8* | Detecto 400 | 50kg | 50 kg | 50 kg |
| 9* | Detecto 400 | 50kg | 49.4 kg | 49.4 kg |

<sup>\*</sup>Scale has not been in field

#### **Number of Measurements Conducted by Scale**

- Cohort 1 baseline height and weight were conducted by UCLA staff using scales 4-6. Scales were not individually labeled.
  - o 236 preschool children and 40 Teachers over 9 sites between 12/05/2019 02/19/2020
- Cohort 1 follow-up/Cohort 2 baseline were conducted by preschool staff using scales #1-6.
  - 362 preschool children and 84 teachers at 26 sites between 10/07/2020 02/26/ 2021

| Cohort 1 Follow-up and Cohort 2 Baseline data collection | | | | |
|---|---|---|---|---|
| Scale Number | Number of Sites | Children weight assessments (n) | Teacher weight assessments (n) | Dates in the Field |
| 1 | 4 | 55 | 16 | 10/16/20 - 1/13/21 |
| 2 | 4 | 61 | 16 | 10/20/20 - 02/19/21 |
| 3 | 6 | 89 | 24 | 10/07/20 - 02/16/21 |
| 4 | 4 | 40 | 12 | 11/05/20 - 02/26/21 |
| 5 | 3 | 40 | 3 | 10/20/20 - 02/26/21 |
| 6 | 5 | 77 | 13 | 10/27/20 - 02/16/21 |
| TOTAL | 26 | 362 | 84 | |

#### Scale summary as of December 2021:

At each assessment, UCLA research staff track scale readings in FORM TO CHECK ACCURACY

In September 2021, UCLA's restrictions on field work lifted; the project returned to the originally planned approach of having UCLA staff members conduct the height and weight measurements.

UCLA Research staff continued to ensure scale accuracy prior to measurement collection. Before height and weight equipment are used in the field, UCLA research staff asses the scales at each of the following calibration weights: 10kg, 20kg, 30kg, 40kg, and 50kg. If the scale is out of calibration at 50kg, the scale was also assessed at 70kg to determine drift (e.g., if a scale read 10kg, 20kg, 30kg, and 40kg accurately, but read 50kg as 49.9kg, the scale was also assessed at 70kg.)

All research scales were in calibration before they were stored in the CPCR office over UCLA's 2021-2022 winter closure.